CLINICAL TRIAL: NCT01829230
Title: Myopia Progression After Ceasing Myopia Control Contact Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-1561AF
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test lens C (Experimental): Test lens C from previous study
  Interventions: Device: 1 Day Acuvue Moist
- Test lens A (Active Comparator): Test lens A from previous study
  Interventions: Device: 1 Day Acuvue Moist

INTERVENTIONS:
Device: 1 Day Acuvue Moist — Lenses will be worn in a daily wear modality

SUMMARY:
This is a continuation study for subjects who were previously fit with test or control lenses; all will stop wearing their study lenses assigned in the previous study and will start to wear an FDA-approved marketed spherical soft contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be enrolled in the parent protocol for at least one year.
2. The subject's parent or legal guardian must read and sign the STATEMENT OF INFORMED CONSENT and the subject must read and sign the Child's Assent Form and be provided a copy of each form.
3. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Ocular or systemic allergies that may interfere with contact lens wear.
2. Systemic disease or autoimmune disease or use of medication (e.g. antihistamine), which may interfere with contact lens wear.
3. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining or any other abnormality of the cornea, which may contraindicate contact lens wear.
4. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection that might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Any infectious disease (e.g. hepatitis, tuberculosis) or an immunosuppressive disease (e.g. HIV)
8. Diabetes
9. Previous refractive surgery, orthokeratology, keratoconus, or other corneal irregularity in either eye. Rigid contact lens wearers cannot be enrolled in the study.
10. Strabismus.
11. Pupil or lid abnormality or infection in either eye
12. Central corneal scar in either eye
13. Aphakia in either eye
14. Contraindications to contact lens wear such as dry eye or history of prior unsuccessful contact lens wear.
15. History of participation in prior clinical trials aimed to control myopia progression, except for the parent trial
16. Surgically altered eyes, ocular infection of any type, ocular inflammation.
17. Anterior chamber angle grade 2 or narrower by Van Herrick method.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Lens C | Test Lens A
Started | 40 | 42
Completed | 39 | 38
Not Completed | 1 | 4
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all randomized subjects in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Lens C | Test Lens A | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 42 | 82
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (1.2) | 11.0 (1.2) | 11.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Axial Length of the Eye
Description: Axial length was measured with the IOLMaster at baseline and then every 6 months throughout the course of the study. Five measurements were collected at each visit from the subject's right eye and the average of the 5 measurements was used for the analysis.
Time Frame: Baseline and every 6 months post-baseline up to 18 months
Population: All subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Groups:
- Test Lens C: Test lens C from the previous study
- Test Lens A: Test lens A from the previous study
Arm/Group | Test Lens C | Test Lens A
Number analyzed (Participants) | 40 | 41
millimeter (mm)
  Change from baseline at 6 months | 0.080 (0.0822) | 0.073 (0.0661)
  Change from baseline at 12 months | 0.229 (0.1237) | 0.231 (0.1181)
  Change from baseline at 18 months | 0.272 (0.1656) | 0.255 (0.1611)

2. Primary Outcome: Spherical Equivalent Refractive Error
Description: Cycloplegic spherical equivalent refraction of the subjects's right eye was computed from the sphero-cylindrical refraction measured with an open-field auto refractor. The median of 5 repeated measurements, each of which was the average of 3 consecutive readings, was used for the analysis.
Time Frame: Baseline and every 6 months up to 18 months
Population: All subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: diopter (D)
Arm/Group | Test Lens C | Test Lens A
Number analyzed (Participants) | 41 | 40
diopter (D)
  Change from baseline at 6 months | -0.015 (0.1911) | -0.155 (0.2101)
  Change from baseline at 12 months | -0.342 (0.3136) | -0.471 (0.2991)
  Change from baseline at 18 months | -0.444 (0.3866) | -0.569 (0.3718)

ADVERSE EVENTS:
Arm/Group | Test Lens C | Test Lens A
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes